CLINICAL TRIAL: NCT06072599
Title: Use of Osteopathic Manipulative Treatment for Non-Musculoskeletal Conditions: A DO-Touch.NET Card Study
Brief Title: Use of Osteopathic Manipulative Treatment for Non-musculoskeletal Conditions
Status: Enrolling by invitation | Type: Observational
Sponsor: A.T. Still University of Health Sciences (Other)
Collaborators: DO-Touch.NET (Unknown)
Responsible Party: Sponsor
Other Study IDs: Non-MSK OMT
Record Dates: First submitted 2023-09-13; First posted 2023-10-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Manipulation, Osteopathic
Keywords: Musculoskeletal Diseases; Non-Musculoskeletal Diseases; Osteopathic Manipulative Treatment
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn how clinicians use osteopathic manipulative treatment (OMT) for their patients who have problems only related to their muscles, bones, and joints (ie, musculoskeletal problems) compared to patients whose problems involve other body systems (eg, infections, breathing, bowel function). The main questions it aims to answer are:

* What percentage of patients receiving OMT have a non-musculoskeletal problem?
* Is there a difference in the OMT techniques when the patient's problems include a non-musculoskeletal problem compared to patients with only musculoskeletal problems?

Surveys will be completed by the clinicians about 20 unique adult (age 18 or older) patients who have received OMT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving osteopathic manipulative treatment from a participating treatment provider

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving osteopathic manipulative treatment globally either in an outpatient or inpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Type of chief complaint | 24 hours
  Multiple choice question: Do this patient's chief complaints include musculoskeletal complaints only, non-musculoskeletal complaints only, or both musculoskeletal and non-musculoskeletal complaints?
Osteopathic manipulative treatment techniques | 24 hours
  Multiple choice question (multiple answers): What OMT techniques did you use to treat this patient's somatic dysfunction? (list of 12 OMT technique categories)

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Johnson, MA, Principal Investigator — A.T. Still University
Locations (1):
- ATSU-KCOM OMM Clinic, Kirksville, Missouri, United States

IPD SHARING:
Plan to Share IPD: No